CLINICAL TRIAL: NCT04850677
Title: Treating Non-typhoidal Salmonella Bloodstream Infections in Children Under Five in DR Congo: a Cohort Study - TreNTS
Brief Title: Treating Non-typhoidal Salmonella Bloodstream Infections in Children Under Five in DR Congo: a Cohort Study
Acronym: TreNTS
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Hôpital St. Luc Kisantu (Unknown); KU Leuven (Other); International Vaccine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ITM202007
Record Dates: First submitted 2021-04-07; First posted 2021-04-20 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Blood-stream Infections; Salmonella Infection Non-Typhoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total: All subjects in the study belong to the same group/cohort. As this is an observational study there is no intervention planned.
  Interventions: Other: Observational Cohort

INTERVENTIONS:
Other: Observational Cohort — Observational study

SUMMARY:
With this study the researchers aim to provide observational data on the treatment efficacy of currently used antibiotic treatment regimens for NTS BSI in hospital-admitted children. The study is an observational cohort study where the antibiotic treatments used and treatment outcomes in the St. Luc general referral hospital in Kisantu health zone (Province Kongo Central, DR Congo) will be described.

DETAILED DESCRIPTION:
In sub-Saharan Africa, non-typhoidal Salmonella (NTS) are a frequent cause of bloodstream infection (BSI) in young children, display high levels of antibiotic resistance and have a high case fatality rate (15%). In Kisantu hospital in the Democratic Republic of Congo (DR Congo), NTS account for 75% of blood culture pathogens in young children.

Currently, NTS BSI are mostly treated with third generation cephalosporins or fluoroquinolones. However, resistance to these antibiotics is emerging in NTS BSI. Third generation cephalosporine and fluoroquinolone resistant Salmonella are identified as critical priority pathogens by the World Health Organization (WHO). To combat the developing antimicrobial resistance, rational and evidence-based antibiotic treatment of NTS BSI is crucial.

So far, there are no guidelines to treat NTS BSI in a low-resource setting. The currently used antibiotic regimens are experience-based or extrapolated from typhoid fever. The absence of dedicated studies addressing antibiotic treatment efficacy in NTS BSI in sub-Saharan African children hampers the development of evidence-based antibiotic treatment guidelines and antibiotic stewardship.

Clinical practice guidelines established for high- and middle-income countries recommend 7 - 14 days of parenteral antibiotic treatment for NTS BSI. In sub-Saharan Africa however, financial, logistic and nursing care barriers preclude such long parenteral treatment regimens.

To decrease the case fatality and combat antibiotic resistance of NTS BSI in its most affected population (i.e. children in sub-Saharan Africa), data that support appropriate antibiotic treatment (i.e. antibiotic class, dose, route and duration) are urgently needed.

The researchers aim to provide observational data on the treatment efficacy of currently used antibiotic treatment regimens for NTS BSI in hospital-admitted children.

They hypothesize that, in terms of treatment efficacy in hospital admitted children with NTS BSI, a short course of parenteral antibiotics (<7 days) with switch to oral antibiotics is not inferior to a full parenteral antibiotic course (≥7 days).

This study is designed as a prospective, single-center, hospital-based observational study on the efficacy of antibiotic treatment of a cohort of young children (1 month to 5 years old) with NTS BSI. Data will be collected from the enrolled children during three different study phases, i.e., upon admission, daily in-hospital follow-up and post-discharge follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Be a child > 28 days and < 5 years old
* Be admitted to Kisantu Hospital
* Have a blood culture sampled upon hospital admission
* Having a caregiver willing and able to provide written informed consent, which will be requested as soon as possible after screening of the other three eligibility criteria. By consenting with study participation of the child, the caregiver agrees to that the child participates in the study procedures at presentation in the hospital, during hospital admission and during 1 month after discharge.

Exclusion Criteria:

* Child died and caregiver left the hospital before enrollment
* Child and caregiver left the hospital before enrollment

Ages: 28 Days to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 28 days and 5 years that are admitted to the Kisantu hospital with a need for a blood sample culture (suspicion of a blood-stream infection).
Sampling Method: Non-Probability Sample
Enrollment: 1884 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Clinical failure (fever) | up to day 7 after start of appropriate antibiotics
  Clinical failure (categorical): composite outcome defined as:
  - the persistence of tympanic temperature > 37.5°C after 7 days of appropriate antibiotic treatment
Clinical failure (death) | from 1st dose of antibiotics until discharge. (maximum period of hospitalization is not defined but is usually maximum 4 weeks)
  Clinical failure (categorical): composite outcome defined as:
  - death between the 1st dose of appropriate antibiotics and discharge

SECONDARY OUTCOMES:
In-hospital survival | from 1st dose of antibiotics until discharge. (maximum period of hospitalization is not defined but is usually maximum 4 weeks)
  In-hospital survival (categorical variable): survival measured between 1st dose of appropriate antibiotics and discharge
Overall survival | One month after discharge (no maximum duration of hospitalization)
  Overall survival (time-to-event): survival time measured between 1st dose appropriate antibiotics and one-month post-discharge
Time to fever clearance | from 1st dose of antibiotics until discharge. (maximum period of hospitalization is not defined but is usually maximum 4 weeks)
  Time to fever clearance (time-to-event): fever clearance is defined as a tympanic temperature ≤37.5°C for at least 2 days [15-17], measured between 1st dose appropriate antibiotics and discharge
Length of hospital stay | from 1st dose of antibiotics until discharge. (maximum period of hospitalization is not defined but is usually maximum 4 weeks)
  Length of hospital stay (time-to-event): number of days that the child was admitted to the hospital, measured between moment of admission and discharge
Microbiological cure | At day 5 of parenteral treatment
  Microbiological cure (categorical): no growth of NTS BSI in the follow-up blood culture taken at the day 5 of parenteral antibiotics
Possible disease recurrence | At one month post-discharge (no maximum period of hospitalization)
  Possible disease recurrence:
  * Fever recurrence: reappearance of objective (measured temperature > 37.5°C) or subjective fever according to the caregiver, measured between moment of fever clearance and one-month post-discharge
  * All-cause hospital readmission: readmission at a hospital or health center irrespective of the cause of readmission, measured between discharge and one-month post-discharge
  * All-cause care seeking at health care facilities: consultation of any health care facility (traditional, private or official) irrespective of the reason for consultation, measured between discharge and one-month post-discharge
  * Re-initiation of antibiotics or antimalarials: start of antibiotic or antimalarial treatment after stop of antibiotic treatment for NTS BSI irrespective of the reason for treatment, measured between last dose of appropriate antibiotics and one-month post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bieke Tack, MD, Principal Investigator — Institute of Tropical Medicine Antwerp
Locations (1):
- Kisantu Hospital, Kisantu, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing procedure for the study will comply with the Institute of Tropical Medicine's data sharing policy on open access to research data. After publishing the manuscript, participant level study data may be shared with other interested users under restricted conditions or made available through an open data repository. These study data will only be shared if the enrolled child are anonymized so that their identity cannot be determined, neither directly nor indirectly. Any subsequent sharing of participant level data will require approval from Institut National de Recherche Biomédicale (INRB) and Institute of Tropical Medicine (ITM).

REFERENCES:
- [Derived] Tack B, Vita D, Mbuyamba J, Ntangu E, Vuvu H, Kahindo I, Ngina J, Luyindula A, Nama N, Mputu T, Im J, Jeon H, Marks F, Toelen J, Lunguya O, Jacobs J, Van Calster B. Developing a clinical prediction model to modify empirical antibiotics for non-typhoidal Salmonella bloodstream infection in children under-five in the Democratic Republic of Congo. BMC Infect Dis. 2025 Jan 27;25(1):122. doi: 10.1186/s12879-024-10319-x. PMID 39871187
- [Derived] Tack B, Vita D, Ntangu E, Ngina J, Mukoko P, Lutumba A, Vangeluwe D, Toelen J, Allegaert K, Lunguya O, Ravinetto R, Jacobs J. Challenges of Antibiotic Formulations and Administration in the Treatment of Bloodstream Infections in Children Under Five Admitted to Kisantu Hospital, Democratic Republic of Congo. Am J Trop Med Hyg. 2023 Oct 30;109(6):1245-1259. doi: 10.4269/ajtmh.23-0322. Print 2023 Dec 6. PMID 37903440